CLINICAL TRIAL: NCT06031038
Title: Impact of Telemonitoring in the Management of Complex Inflammatory Bowel Disease in Spain: TECCU Multicenter Study
Brief Title: Impact of Telemonitoring in the Management of Complex IBD in Spain: M-TECCU
Acronym: M-TECCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M-TECCU
Record Dates: First submitted 2023-07-24; First posted 2023-09-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Telemedicine
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: To compare the time in remission of patients with complex IBD (require immunosuppressants and/or biologics to control their luminal inflammatory activity) controlled with the TECCU intervention (G_TECCU) with respect to usual clinical practice (G_Control) after 52 weeks of follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients receive conventional care in the outpatient clinics of the participating specialized IBD units in Spain. This is complemented with telephone controls for those aspects that can be controlled by this means according to standard clinical practice. Likewise, an individual assessment will be made if, after the situation generated by SARS-COV2, any participating center should have to modify face-to-face consultations for telephone consultations, following the usual clinical practice at all times.
- Web telemonitoring group (G_TECCU) (Active Comparator): Monitoring and control will be done remotely through the TECCU comprehensive management platform, configured to respond to the specific needs of IBD patients. Patients will connect to the internet from a computer or an APP application on a tablet or mobile terminal, Android or iOS. They will have to complete questionnaires related to the variables under study at each control according to a pre-established follow-up plan. During the follow-up, the number of controls may be increased (intensive monitoring) according to the evolution of the patient, who in turn will be able to perform controls on demand. The healthcare personnel of each IBD unit will receive the information of each patient filtered through an intelligent alert generation system from which an integrated intervention protocol will be followed to adjust the treatment and follow-up plan in each case.
  Interventions: Other: TECCU Software

INTERVENTIONS:
Other: TECCU Software — patient monitoring by software application
  Arms: Web telemonitoring group (G_TECCU)

SUMMARY:
M-TECCU is a study: multicenter, randomized and open. It consists of two parallel groups to compare the efficacy of the TECCU web-based telemonitoring system to achieve and maintain activity remission in patients with moderate-high complexity inflammatory bowel disease compared to usual clinical practice.

DETAILED DESCRIPTION:
Clinical trial with an open, randomized and controlled non-inferiority medical device, in which the impact of a follow-up method through a web telemonitoring platform on the time in clinical remission of patients with complex IBD is evaluated, in comparison with the usual follow-up in outpatient clinics.

Patients with complex IBD are considered to be those who receive treatment with immunosuppressants or biological therapies to control the luminal activity of their disease. Patients carry out periodic controls for the disease according to a pre-established schedule based on national and international clinical guidelines. The patients in the telemonitoring group (G_TECCU) follow these controls through the TECCU platform, a web system that allows them to fill in questionnaires related to the clinical variables under study and communicate freely with healthcare personnel during pre-established controls and when the patient deems it necessary. On the other hand, the patients of the control group (G_Control) carry out the controls according to the same schedule as G_TECCU, but following the usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18a
* IBD (CD or UC) diagnosed according to ECCO criteria
* Start treatment with immunosuppressants and/or biological therapies due to luminal activity
* signed informed consent

Exclusion Criteria:

* Pregnant women
* Presence of active perianal disease, ileoanal reservoir, or definitive stoma
* Patients with mental illness or other poorly controlled illness
* Patients with active cancer diagnosis
* Terminal patients and/or palliative care (SECPAL)
* Family members of the research team
* Patients without a telephone line to connect with a mobile, tablet and/or computer / Inability to drive
* Cognitive or linguistic difficulties
* Patients included in another experimental study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
clinical remission | 52 weeks
  To compare the time in remission of patients with complex IBD (require immunosuppressants and/or biologics to control their luminal inflammatory activity) controlled with the TECCU intervention (G_TECCU) with respect to usual clinical practice (G_Control) after 52 weeks of follow-up.

SECONDARY OUTCOMES:
cost-effectiveness | 52 weeks
  Carry out a cost-effectiveness analysis based on the direct and indirect costs generated during the 12-month follow-up in G_TECCU and G_control.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Aguas, Principal Investigator — Spanish Working Group on Crohn's disease and ulcerative colitis (GETECCU)
Locations (30):
- Spain (30):
  - Hospital Universitario y Politécnico la Fe, Valencia, Valencia
  - Hospital Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Cabueñes, Cabueñes
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital de Cruces, Cruces
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Trueta de Girona, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital de Huelva, Huelva
  - Hospital Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Puerta del Hierro, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital de Manresa, Manresa
  - Hospital Morales Meseguer, Murcia
  - Hospital Parc Taulí de Sabadell, Sabadell
  - Hospital Infanta Sofía, San Sebastián de los Reyes
  - Hospital Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario de Santiago, Santiago de Compostela
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Universitario Mutua Terrassa, Terrassa
  - Hospital Clínico Universitario Valencia, Valencia
  - Hospital de Vigo, Vigo
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miquel Servet, Zaragoza

REFERENCES:
- [Background] Del Hoyo J, Nos P, Faubel R, Munoz D, Dominguez D, Bastida G, Valdivieso B, Correcher M, Aguas M. A Web-Based Telemanagement System for Improving Disease Activity and Quality of Life in Patients With Complex Inflammatory Bowel Disease: Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Nov 27;20(11):e11602. doi: 10.2196/11602. PMID 30482739
- [Background] Aguas M, Del Hoyo J, Faubel R, Munoz D, Dominguez D, Bastida G, Navarro B, Barrios A, Valdivieso B, Correcher M, Nos P. A Web-Based Telemanagement System for Patients With Complex Inflammatory Bowel Disease: Protocol for a Randomized Controlled Clinical Trial. JMIR Res Protoc. 2018 Dec 21;7(12):e190. doi: 10.2196/resprot.9639. PMID 30578197
- [Background] Del Hoyo J, Aguas M. Cost-effectiveness of Telemedicine-directed Specialized vs Standard Care for Patients With Inflammatory Bowel Diseases in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Jan;19(1):206-207. doi: 10.1016/j.cgh.2020.06.016. No abstract available. PMID 33339564
- [Derived] Aguas M, Del Hoyo J, Vicente R, Barreiro-de Acosta M, Melcarne L, Hernandez-Camba A, Madero L, Arroyo MT, Sicilia B, Chaparro M, Martin-Arranz MD, Pajares R, Mesonero F, Manosa M, Martinez P, Chacon S, Tosca J, Marin S, Sanroman L, Calvo M, Monfort D, Saiz E, Zabana Y, Guerra I, Varela P, Baydal V, Faubel R, Corsino P, Porto-Silva S, Brunet E, Gonzalez M, Gutierrez A, Nos P. Telemonitoring of Active Inflammatory Bowel Disease Using the App TECCU: Short-Term Results of a Multicenter Trial of GETECCU. J Med Internet Res. 2024 Nov 18;26:e60966. doi: 10.2196/60966. PMID 39189160